CLINICAL TRIAL: NCT07386067
Title: Mesh Design for Open Inguinal Hernia Repair: Superior Outcomes and Fewer Complications
Brief Title: Mesh Design for Open Inguinal Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Yasser Ali Orban, assisstant professor, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mesh Design
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Mesh; Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hernia arm represent patients with inguinal hernia (Experimental): the new mesh desined to fit the posterior wall of inguinal canal
  Interventions: Procedure: new mesh design for inguinal hernia

INTERVENTIONS:
Procedure: new mesh design for inguinal hernia — the new mesh design is cut to fit the posterior wall of the inguinal canal

SUMMARY:
Inguinal hernia repair is the most common operation performed by general surgeons worldwide, surgical repair is the only established definitive treatment for inguinal hernia with multiple variable described approaches, Since Lichtenstein and his colleagues pronounced the use of mesh in tension-free inguinal hernia repair, the open Lichtenstein mesh repair of inguinal hernia became a standard of care for inguinal hernia repair due to easiness of performance with low recurrence rates (1, 2, 3).

In the past many different factors have been identified to reduce chronic postoperative inguinal pain CPIP, Sophisticated studies suggested that mechanical mesh fixation should be avoided, and proper knowledge of inguinal nerves is essential (4-9).

Surgeons must consider patient characteristics and mesh properties when selecting a mesh for hernia treatment. Mechanical compatibility between meshes and abdominal wall layers is crucial for avoiding complications. Lightweight, monofilament meshes with large pores and minimal surface area are ideal; however, the surgeon should never forget that the way the mesh is positioned as important as the type of mesh used. Despite the new materials available, surgical skill still has a major role in preventing hernia post-operative complications and recurrence. Future research will continue to focus on the surgical techniques and biomaterials to achieve the best outcomes (10).

Our method uses a smaller single mesh that covers all weaknesses in the inguinal canal and is covered with a fibro-cremasteric sheath to prevent the prosthesis from coming into touch with neural processes. This method is applicable to all cases of primary inguinal hernia.

ELIGIBILITY:
Inclusion Criteria:

* • males older than 18 years old with primary inguinal hernia.

Exclusion Criteria:

* females patients with bleeding tendency.

  * Complicated inguinal hernia.
  * Huge inguinoscrotal hernia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
hernia recurrence | 6 months following the operation
  The rate of return of the hernia in the same location.

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig Univeesity Hospitals, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No